CLINICAL TRIAL: NCT01354392
Title: A Phase 2 Trial of AZD1152 in Relapsed/Refractory Diffuse Large B-cell Lymphoma
Brief Title: AZD1152 in Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: The Christie NHS Foundation Trust (Other); University of Manchester (Other); Early Phase Cancer Research Hub, Oxford (Unknown)
Responsible Party: Principal Investigator, Linda Ward, QA Coordinator, Cancer Centre, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORH/PID/6265
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Lymphoma
Keywords: Relapsed or refractory; Large B-Cell; Diffuse
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — 2-((3-((4-((5-(2-((3-fluorophenyl)amino)-2-oxoethyl)-1H-pyrazol-3-yl)amino)quinazolin-7-yl)oxy)propyl)(ethyl)amino)ethyl dihydrogen phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD1152 (Experimental)
  Interventions: Drug: AZD1152

INTERVENTIONS:
Drug: AZD1152 — Up to 6 cycles. Each cycle consists of 800 mg. IV infusion over 96 hrs.

SUMMARY:
Diffuse large B-cell lymphoma is the commonest type of aggressive non-Hodgkin's lymphoma, a type of cancer of a cell called a lymphocyte which makes up part of the immune system. Although most patients are cured with chemotherapy used as initial treatment, about 20-30% of patients still experience relapse. Curing relapsed disease is much less successful, even with the use of high doses of chemotherapy and stem cell transplant. There is then an urgent need for effective, new agents to treat patients with diffuse large B-cell lymphoma who have relapsed or who have developed resistance to other forms of chemotherapy.

This trial is using a drug called AZD1152 which interferes with the ability of a cancer cell to divide and grow. It has been used before in patients with other types of cancer, but never before in lymphoma patients. Responses in other cancers have been seen, particularly in leukaemia which is a disease related to lymphoma. The investigators are planning to use this agent in 15 patients with diffuse large B-cell lymphoma in which potentially curative treatments have failed. The main aim is to see whether the drug shows any activity in this type of lymphoma. This will be mainly assessed using CT and PET scans. The investigators are also investigating how well a blood test can predict both the response to the drug and the toxicity of the drug - this is called a biomarker study and forms part of the clinical trial. The other main aim of the study is to assess the toxicity of the treatment. Previous studies in humans suggest the drug is reasonably well tolerated, although side effects such as stomatitis (soreness of the mouth) and suppression of the bone marrow (leading to risk of infection and bleeding) have been seen.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged ≥ 18 yrs.
* ECOG performance score of 0, 1 or 2.
* Life expectancy of at least 12 weeks.
* Haematological and biochemical indices within the ranges shown below Lab Test Value required Haemoglobin (Hb) ≥ 9g/dL White Blood Count (WBC) ≥ 2x109/L Platelet count ≥ 100x109/L Absolute Neutrophil count ≥ 1.0x109/L; Serum bilirubin ≤ 1.5 x ULN AST (SGOT) or ALT ≤ 1.5 x ULN Creatinine clearance (Cockcroft-Gault) > 50 ml/min
* Relapsed or refractory DLBCL in which all participants must have received at least one potentially curative established immunochemotherapy lymphoma regimen that contained rituximab (e.g. R-CHOP, R-PMitCEBO, R-GCVP, R-CNOP). Participants must also have failed or be ineligible for salvage/high dose therapy.
* Relapsed or refractory DLBCL proven by biopsy (within 6 months of enrolment in trial); either de novo DLBCL or transformed follicular lymphoma.
* At least 1 lesion (> 1.5cm), not previously irradiated, that can be accurately measured on CT and which is FDG avid on CT-PET scanning, as defined by Cheson criteria.
* Able to give informed consent and capable of co-operating with protocol.

Exclusion Criteria:

* Any anti-cancer therapy (including radiotherapy and participation in other clinical trials) within 28 days prior to Day 1. Patients may however be receiving corticosteroids as an anti-lymphoma treatment of 50mg daily prednisolone or equivalent up until screening. At screening (or before) this must be tapered down so that they are only on a low dose (10mg daily or less) by the time AZD1152 commences. This may be continued for indications other than lymphoma treatment throughout the study.
* Any unresolved toxicity from prior anti-cancer therapy greater than CTCAE grade I (except alopecia).
* Previous treatment with aurora kinase inhibitors.
* Clinical evidence of central nervous system involvement.
* Another active malignancy within the past five years, except adequately treated basal or squamous cell carcinoma of the skin, or carcinoma of the cervix in situ.
* Clinically significant and uncontrolled major medical condition(s) including but not limited to: active infection, bleeding diathesis, symptomatic congestive heart failure, cardiac arrhythmia or psychiatric illness/social situations which would limit compliance with protocol requirements.
* Major surgery within 4 weeks prior to entry into the study (excluding placement of vascular access or biopsy) that involved general anaesthesia or respiratory assistance.
* Mean QTc interval > 470 ms calculated from 3 ECGs using Fridericia's or Bazett's correction on 12-lead ECG machine.
* Serologically positive for HIV, hepatitis B or C assessed within 28 days of initiation of study treatment using an ELISA method performed by an HPA accredited laboratory.
* Participants of reproductive potential not willing to use adequate contraceptive measures for the duration of the study (both male and female participants).
* Pregnant or breastfeeding women. Female participants must have a negative urinary or serum pregnancy test when done or have evidence of post-menopausal status (Defined as absence of menstruation for greater than 12 months, bilateral oophorectomy or hysterectomy).
* Participants who have had live attenuated or yellow fever vaccines within 6 months of trial beginning.
* Participants not willing and able to comply with the protocol for the duration of the study, and scheduled follow-up visits and examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR; Cheson 2007 criteria) | ORR will be calculated from the data obtained from the End Visit, which occurs approx. 14 days after the end of the last cycle of treatment the patient undergoes.

SECONDARY OUTCOMES:
Progression free survival at 1 year | PFS will be calculated at some point 1-year post-study from the available 1 year post-study data.
Percentage change in tumour size | Percentage change in tumour size will be calculated from the data obtained from the End Visit, which occurs approx. 14 days after the end of the last cycle of treatment the patient undergoes.
Safety of AZD1152 | The safety of AZD1152 is monitored at every study visit on study via recording AEs/SAEs/SUSARs. However, these are also recorded as they arise. E.g. they would be recorded if the patient had an emergency admissions.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Hatton, MRCPath FRCPath(UK) MRCP FRCP, Study Director — Oxford Radcliffe NHS Trust & University of Oxford; John A Radford, MB, ChB, MRCP, MD, FRCP, Principal Investigator — University of Manchester, Christie NHS Foundation Trust; Graham P Collins, MBBS, MRCP(UK), FRCPath, Principal Investigator — Oxford Radcliffe NHS Trust, University of Oxford
Locations (2):
- United Kingdom (2):
  - Christie NHS Foundation Trust (Christie Hospital), Machester, Lancashire
  - Oxford Radcliffe NHS Trust (Cancer & Haematology Centre, Churchill Hospital), Oxford, Oxfordshire

REFERENCES:
- [Derived] Collins GP, Eyre TA, Linton KM, Radford J, Vallance GD, Soilleux E, Hatton C. A phase II trial of AZD1152 in relapsed/refractory diffuse large B-cell lymphoma. Br J Haematol. 2015 Sep;170(6):886-90. doi: 10.1111/bjh.13333. Epub 2015 Feb 26. No abstract available. PMID 25721307